CLINICAL TRIAL: NCT02882373
Title: L-Arginine For Anti-VEGF Induced Kidney Injury
Brief Title: Arginine in Treating Patients With Anti-VEGF Induced Kidney Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator's Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-1105; NCI-2018-02537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-1105 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-08-22; First posted 2016-08-29 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Drug-Induced Nephropathy; Hypertension; Proteinuria
MeSH Terms: conditions — Hypertension; Proteinuria | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (arginine) (Experimental): Patients receive arginine PO QID. Treatment continues for up to 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Arginine
- Group II (placebo) (Placebo Comparator): Patience receive placebo PO QID. Treatment continues for up to 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Arginine — Given PO
  Other Names: Amino-5-guanidino-pentanoic acid; Arg; L-Arginine
  Arms: Group I (arginine)
Drug: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)

SUMMARY:
This phase II trial studies how well arginine works in treating patients with kidney injury caused by anti-VEGF drugs used in standard treatment for cancer. Arginine is a nutritional supplement that may control side effects of anti-cancer drugs such as high blood pressure and protein in the urine and may also help to improve kidney function in patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the value and/or limitations of using orally supplemented arginine (L-arginine) to improve renal function associated with the use of anti-angiogenic therapies that target vascular endothelial growth factor (VEGF).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive arginine orally (PO) four times daily (QID). Treatment continues for up to 3 months in the absence of disease progression or unacceptable toxicity.

GROUP II: Patience receive placebo PO QID. Treatment continues for up to 3 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up within 1 month.

ELIGIBILITY:
Inclusion Criteria:

* On or enrolled for anti-VEGF therapy
* Systolic Blood Pressure >= 140 mm Hg
* Diastolic Blood Pressure >= 90 mm Hg
* Proteinuria >= 500 mg/day or worsening glomerular filtration rate (GFR) (> 0.3 mg/dl in 48 hours [hrs.] or > 50% decline from baseline creatinine in 1 week)

Exclusion Criteria:

* Allergy to L-arginine
* Systolic Blood Pressure < 140 mm Hg
* Diastolic Blood Pressure < 90 mm Hg
* Proteinuria < 500 mg/day
* Continuous tube feeds (since the medication will be given in-between meals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Reduction in proteinuria as measured by protein-creatinine ratio (UPC) > 500 mg/day | Baseline up to 3 months
  Linear mixed effects regression will be utilized to analyze the longitudinal change of UPC between treatment and placebo groups.

SECONDARY OUTCOMES:
Improved glomerular filtration rate (GFR) >= 25% | Baseline up to 3 months
  Linear mixed effects regression will be utilized to analyze the GFR between treatment and placebo groups.
Reduction in systolic blood pressure (SBP) >= 10 mmHg and/or diastolic blood pressure >= 5 mmHg | Baseline up to 3 months
  Linear mixed effects regression will be utilized to analyze the SBP between treatment and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Danesh, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States